CLINICAL TRIAL: NCT01169441
Title: EXTRACT Study (Data Collection on the Extraction of 2nd and 3rd Generation Defibrillation Leads)
Brief Title: Lead Extract Study
Acronym: EXTRACT
Status: Completed | Type: Observational
Sponsor: St. Paul Heart Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Pierce Vatterott, MD, St. Paul Heart Clinic
Other Study IDs: #2265-4
Record Dates: First submitted 2009-05-28; First posted 2010-07-26 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2009-05

CONDITIONS: Cardiac Surgical Procedures
Keywords: ICD leads; Removal; Extraction; Ventricular leads; Extract; laser; Observe the lead with x-ray during movement and collect information on current ways of removing an ICD lead.

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The recent expansion of indications for implantable cardioverter defibrillators (ICDs) has changed the population of patients being implanted. Younger and healthier patients are now being implanted for primary prevention of sudden cardiac death. Due to the younger population, the likelihood of the lead failing during the lifetime of the patient is higher and also more likely to need extraction. To reduce the risk of the lead extraction procedure and therefore reduce the number of abandon leads, ICD lead manufacturers are designing leads to offer improved chronic extractability to reduce the morbidity and mortality during these procedures.

DETAILED DESCRIPTION:
This study will enroll up to 100 subjects at our site only. Prior to the procedure information will be collected including the subjects demographics, medications, medical, cardiovascular and surgical history. During the lead extraction procedure specific data will be gathered which includes items such as: total lead length, lead length from insertion site to connector end of lead just prior to lead extraction, extraction tools used and the physician description of the extraction. The patients will undergo an assessment of extraction force up to 3 kilograms maximum to the ICD lead for a specified amount of time before the use of laser or extraction sheaths. Extraction forces and approximate times will be monitored and recorded throughout the procedure. Forces will be measured by using a force gauge. Xrays will be taken to show lead position during movement of the arm at the side, above the head and across the chest. Fluoroscopy images of the heart may be saved. The amount of extra time added to the case in order to perform this study and collect the data is estimated at 10 minutes. Participation in the study is complete following the procedure. There is a 30-day follow-up phone call to capture any adverse events which require a clinic visit, ER visit or hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older,
* be scheduled for an ICD lead extraction and
* willing and able to sign the informed consent.

Exclusion Criteria:

* Patients with lead implant duration less than 6 months,
* patients with gross chronic lead infections,
* patients with epicardial or subcutaneous ICD systems (without transvenous ICD lead) and
* patients who are pregnant or suspect they may be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled for an ICD lead extraction
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierce J. Vatterott, M.D., Principal Investigator — St. Paul Heart Clinic
Locations (1):
- St. Paul Heart Clinic, Saint Paul, Minnesota, United States